CLINICAL TRIAL: NCT02180542
Title: Atrial Fibrillation and Premature Atrial Complexes in Patients With Ischemic Stroke: Prevalence, Characteristics and Prognosis
Brief Title: Atrial Fibrillation and Premature Atrial Complexes in Patients With Ischemic Stroke.
Acronym: Pacific
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kristina Hoeg Vinther, Medical Doctor, Odense University Hospital
Other Study IDs: Pacific
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Stroke; Atrial Fibrillation; Premature Atrial Complexes
Keywords: stroke; Ischemic stroke; Cerebral infarction; recurrent stroke; atrial fibrillation; premature atrial complexes; heart rhythm monitoring; left atrial function; carotid artery; plaque morphology
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Atrial Premature Complexes; Ischemic Stroke; Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ischemic stroke patients: Patients admitted with ischemic stroke from march 2012 to april 2014

SUMMARY:
The purpose of this study is to improve secondary prevention of ischemic stroke patients by

1. Estimating prevalence and the prognostic significance of frequent premature atrial complexes in ischemic stroke patients in relation to death, recurrent stroke and atrial fibrillation.
2. Characterize ischemic stroke patients by

   1. Echocardiographic characteristics
   2. Biochemical markers
   3. Plaque composition in the carotid arteries

      * in order to improve risk stratification.

DETAILED DESCRIPTION:
Patients with atrial fibrillation (AF) have a five-fold increased risk of ischemic stroke compared to the general population. Identifying AF can be challenging, but prolonged rhythm monitoring of ischemic stroke patients have shown to enhance detection rates of AF. Therefore it is important to identify predictors of AF to allow targeted screening of patients after ischemic stroke and thereby reduce the recurrent stroke rate. Few former studies have shown an association between excessive numbers of premature atrial complexes (PACs) and AF.

The study population of ischemic stroke patients will at admission undergo following examinations:

1. ECG
2. 48 hours inpatient cardiac telemetry (If not known AF)
3. 24 hours holter monitoring (if not known AF)
4. echocardiogram
5. blood sample
6. CT scan of carotid arteries with contrast made on Dual Energy CT scan.

In the follow-up period, patients will have two visits with 48 hour holter monitoring (after 6 and 12 months, respectively) It will be noticed if patients have any recurrent events, die og developing AF.

The study population will be divided into four groups as follows:

1. patients with new AF at admission
2. patients with known AF
3. patients with frequent PACs
4. patients without frequent PACs. These groups will be compared on baseline characteristics and on outcome as mentioned.

The overall perspective is to make better strategies for detecting occult AF after ischemic stroke to improve secondary stroke prevention care.

ELIGIBILITY:
Inclusion Criteria:

* admitted with ischemic stroke at a single center
* time from diagnose to inclusion maximum 7 days.
* written informed consent or surrogate informed consent eligible
* age > 18 years.

Exclusion Criteria:

* hemorrhagic stroke
* terminal illness and expected lifespan of less than 6 months.
* any physical or mental condition which make the patients unsuitable for participation in the study.
* known with a pacemaker
* anticoagulation treatment of other reasons than atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients admitted to the hospital
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
time to death and recurrent stroke | Up to 4 years

SECONDARY OUTCOMES:
Time to death, recurrent stroke and atrial fibrillation | Up to 4 years
Left atrial volume and function estimated by echocardiography | baseline
  descriptive comparison in between groups.

OTHER OUTCOMES:
biochemical markers | baseline
  descriptive comparison in between groups
Plaque analysis i the carotid arteries on CT | baseline
  descriptive comparison in between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina H Vinther, MD, Principal Investigator
Locations (1):
- Department of Medical Research, OUH, Svendborg, Svendborg, Funen, Denmark